CLINICAL TRIAL: NCT00636519
Title: Botulism Antitoxin Effects on Paralysis Induced by Type A and Type B Botulinum Neurotoxins in the Extensor Digitorum Brevis Muscle
Brief Title: Botulism Antitoxin Effects on Paralysis Induced by Botulinum Neurotoxins in the EDB Muscle
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emergent BioSolutions (Industry)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BT002
Record Dates: First submitted 2008-03-11; First posted 2008-03-14 (Estimated); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Healthy Volunteers
Keywords: Botulism Antitoxin,Heptavalent,Bivalent,EDB Muscle,Paralysis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Stage A (Experimental): Botulism Antitoxin Bivalent (Equine) Types A and B Vs. Placebo
  Interventions: Biological: Botulism Antitoxin Bivalent (Equine) Types A and B
- Stage B (Experimental): Botulism Antitoxin Heptavalent (Equine) Types A-G Vs. Placebo
  Interventions: Biological: Botulism Antitoxin Heptavalent (Equine) Types A-G

INTERVENTIONS:
Biological: Botulism Antitoxin Bivalent (Equine) Types A and B — One vial of Botulism Antitoxin Bivalent(Equine) Types A and B (1:10 in saline) or an Equivalent Volume of Placebo on Day 0 in Stage A
  Arms: Stage A
Biological: Botulism Antitoxin Heptavalent (Equine) Types A-G — One vial of Heptavalent Botulism Antitoxin (1:10 in saline) or an Equivalent Volume of Placebo on Day 0 in Stage B
  Arms: Stage B

SUMMARY:
The primary purpose of this study is:

1. To evaluate the model determined by the ability of botulism antitoxin (bivalent, Aventis) to neutralize Botulinum toxin in the Extensor Digitorum Brevis model of muscle paralysis in Stage A.
2. To assess the ability of botulism antitoxin (heptavalent, Cangene) to neutralize Botulinum toxin in the Extensor Digitorum Brevis model of muscle paralysis in Stage B.

DETAILED DESCRIPTION:
Botulism is a rare disease; however Botulinum toxins (neurotoxins) may be used as biological weapon especially in the form of aerosol. Botulism is caused by neurotoxins that are produced by the obligate anaerobic, gram-positive, spore-forming bacterium Clostridium botulinum (1). C. botulinum produces 8 serologically distinct neurotoxins identified as serotypes A, B, C1, C2, D, E, F, and G (2).

Therapy for botulism includes supportive care and passive immunization with antitoxin. Antitoxin should be administered to patients with neurologic signs of botulism as soon as possible after clinical diagnosis (3). Botulism antitoxin is prepared from plasma obtained from horses that have been immunized with a specific subtype of botulism toxoid and toxin.

The BT-002 is an exploratory pharmacodynamic study that is being performed to evaluate the effect of Botulism Antitoxins in preventing paralysis of extensor digitorum brevis muscle following BOTOX®/ MYOBLOC® administration. This study will compare bivalent and heptavalent products to a placebo. Safety data will be collected.

NP-018 (heptavalent equine-derived botulinum antitoxin) is prepared from plasma obtained from horses that have been immunized with a specific subtype of botulinum toxoid and toxin. Each individual horse is immunized against a single botulinum toxin subtype. Plasma is pooled from horses that have been immunized with the same botulinum toxin subtype. For each antitoxin serotype (A-G), a despeciated product will be produced by pepsin digestion of the IgG monomer in the equine plasma, yielding predominantly F(ab')2 fragment. Following the formulation, the seven antitoxin serotypes will be blended into a heptavalent product and filled into single-use vials. '

This research study will be conducted in two stages - Stage A and Stage B. If enrolled in the Stage A of the study, the subject will have an equal chance of getting either bivalent botulism antitoxin or placebo. If enrolled in Stage B of the study, the subject will have an equal chance of getting heptavalent botulism antitoxin (NP-018) or placebo. The subject will be receiving injections of Botox and Myobloc on the next day after the antitoxin administration in the left and right foot respectively. The subject's participation in this study will be for maximum of 57 days.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 - 55 years
* Body-mass index 19-30
* Normal and healthy as determined by medical history, physical examination, ECG, NCS, vital signs and tests of liver, kidney and hematological functions
* Adequate form of contraception for female subjects

  * For women with child-bearing potential-using hormonal contraception (oral, injectable or implant) continuously for 3 months prior to the start of the study and willing to continue to use hormonal contraception throughout the entire study. IUD inserted or use of condoms for at least 2 months prior to dosing
  * Other forms of contraception may be considered as adequate at physician's discretion
  * Surgically-sterilized female subjects
  * For female subjects who are postmenopausal, an FSH ≥ than 40 mIU/mL must be obtained. If the FSH is < 40 mIU/mL the subject must agree to use an acceptable form of contraception (see above for acceptable forms of contraception)
* Signed written Informed Consent

Exclusion Criteria:

* Previously injected with BOTOX®, BOTOX® COSMETIC or MYOBLOC®
* Any known or documented Botulinum infection/intoxication
* Any known or documented allergies to horses (e.g. rash, wheezing, rhinitis etc. after exposure to horses)
* Any known or documented allergies to horse serum (observation of adverse events after treatment with any kind of product containing horse serum)
* Any moderate or severe food allergies, seasonal allergies or hay fever requiring treatment with peroral or parenteral immunosuppressive drug
* Any known or documented hypersensitivity to blood products derived from a human or equine source
* Any known or documented hypersensitivity to albumin
* Positive result for Botulism Antitoxin skin sensitivity testing
* Any known or documented allergy to rubber, latex or plastic
* Known acute or chronic moderate or severe asthma requiring treatment with peroral and / or parenteral immunosuppressive drugs
* Previously diagnosed or currently suspected Multiple Sclerosis or other neuromuscular degenerative disorder
* Previously diagnosed or currently suspected motor neuron disease
* Previously or currently diagnosed peripheral neuropathy of lower extremities' nerves
* Current infection of the skin / skin problems at the injection site (foot)
* Scar tissue or tattoo of the skin over the extensor digitorum brevis muscles.
* Previously diagnosed or currently suspected diabetes
* Previously diagnosed or currently suspected coagulopathies
* Previously diagnosed or currently suspected vasculitis
* Current treatment or treatment in the past 7 days with aminoglycosides, clindamycin, quinolines or aminopyridine
* Heavy smokers (>10 cigarettes/day)
* History of, or suspected substance abuse (including alcohol) or failure of drug screen at screening or at baseline
* Use of any investigational product within the past 30 days (prior to screening)
* Pregnancy or lactation
* Positive serological test for diagnosis of HIV infection, HBV hepatitis, or HCV hepatitis
* Abnormal (based on principle investigator assessment) nerve conduction study (NCS) results

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2008-02; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Nerve Conduction Study | Screening, Baseline (Day 0, -3 hrs), Day 1 (-1 hr), Day 3, Day 4, Day 7, Day 14, Day 21, Day 28 or Early Withdrawal

SECONDARY OUTCOMES:
Hematology | Screening, Baseline (Day 0, -3 hr), Day 7, Day 14, Day 21, Day 28 or Early Withdrawal
Blood Chemistry | Screening, Baseline (Day 0, -3 hr), Day 7, Day 14, Day 21, Day 28 or Early Withdrawal
Urinalysis | Screening, Baseline (Day 0, -3 hr), Day 7, Day 14, Day 21, Day 28 or Early Withdrawal
Serum anti-Botulism Antitoxin Reactivity | Baseline, Day 28 or Early Withdrawal
Adverse Events | Day 0, Day 1( -1 hr), Day 1, Day 3, Day 4, Day 7, Day 14, Day 21, and Day 28 or Early Withdrawal
Vital Signs | Screening, Day 0 (-3 hrs), Day 0, Day 1 (-1 hr), Day 1, Day 3, Day 4, Day 7, Day 14, Day 21, and Day 28 or Early Withdrawal
Physical Examination | Screening, Baseline (Day 0, -3 hrs), Day 1 (-1 hr), Day 3, Day 4, Day 7, Day 21 and Day 28 or Early Withdrawal
12-lead ECG | Screening/ Day 28 or Early Withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Richard Sloop, M. D., Principal Investigator — R. Richard Sloop, M. D.; Gordon Peterson, Dr., Principal Investigator — Faculty Physicains & Surgeons of Loma Linda University School of Medicine, Department of Neurology
Locations (2):
- United States (2):
  - Dr. Gordon Peterson, Loma Linda, California
  - R. Richard Sloop, M. D., Yakima, Washington

REFERENCES:
- [Background] Benedetto AV. The cosmetic uses of Botulinum toxin type A. Int J Dermatol. 1999 Sep;38(9):641-55. doi: 10.1046/j.1365-4362.1999.00722.x. No abstract available. PMID 10517680
- [Background] Carruthers A, Carruthers J. Cosmetic uses of botulinum A exotoxin. Adv Dermatol. 1997;12:325-47; discussion 348. No abstract available. PMID 8973746
- [Background] Tacket CO, Shandera WX, Mann JM, Hargrett NT, Blake PA. Equine antitoxin use and other factors that predict outcome in type A foodborne botulism. Am J Med. 1984 May;76(5):794-8. doi: 10.1016/0002-9343(84)90988-4. PMID 6720725